CLINICAL TRIAL: NCT00509834
Title: A Phase-IIa, Double-blind, Randomized Study on the Tolerability and Early Efficacy of hLF1-11 in Hospitalized Patients With Proven Candidaemia. (SLIC: Study of Lactoferrin Peptide in Infections With Candida)
Brief Title: A Study on the Tolerability and Early Efficacy of hLF1-11 in Patients With Proven Candidaemia
Acronym: SLIC
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Patient population not available
Sponsor: AM-Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMP IC 01-01
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2008-04

CONDITIONS: Candidaemia
Keywords: hLF1-11; Candida; candidaemia; lactoferrin
MeSH Terms: conditions — Candidemia; Torulopsis | interventions — lactoferrin (1-11), human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hLF1-11 (Experimental): hLF1-11 0.5mg
  Interventions: Drug: hLF1-11
- Placebo (Placebo Comparator): Placebo formulation is Similar to hLF1-11 iv formulation except for the active component
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: hLF1-11 — The study treatment consists of IV administration of:
  (A) hLF1-11 (0.5mg IV bolus daily for 14 days) + fluconazole (up to 1g IV four times daily; 14 days): Group #1, n=10; OR (B) Fluconazole (up to 1g IV four times daily; 14 days) + matching placebo for hLF1-11: Group #2, n=10
  Arms: hLF1-11
Drug: hLF1-11 — 0.5mg hLF1-11 iv per day for 14 consecutive days
  Other Names: human lactoferrin 1-11
  Arms: hLF1-11
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a phase-I, double-blind, randomized study with hLF1-11 to study the tolerability and early efficacy of hLF1-11 compared to standard fluconazole therapy in hospitalized patients with invasive Candida infection.

DETAILED DESCRIPTION:
RATIONALE FOR THE STUDY

Choice of Drug

Fluconazole is considered "standard care" for the treatment of Candida infections, including candidaemia in hospitalized patients.

Preclinical data has demonstrated that hLF1-11 possesses potent antimycotic effects against Candida sp and, importantly, to be synergistic with fluconazole, whereby Candida strains that are fluconazole-resistant become sensitive through the addition of hLF1-11

Choice of Patient Population

Based on preclinical data hLF1-11 has been shown to possess potent effects on Candida albicans models in vitro and in vivo. Furthermore, candidaemia (bloodstream Candida infection) is one of the most likely settings to elicit a therapeutic response since the product is presented as an intravenous formulation

As previously mentioned, fluconazole and hLF1-11 exhibit a synergistic effect in preclinical studies, whereby the effect of fluconazole is enhanced by the addition of hLF1-11.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before admission in the study.
* Patients in whom Candida species have been confirmed by 2 consecutive blood cultures within 12 hours.
* Patients who have not received systemic administration of antifungal agents or who have started such administration within 48 hours prior to entry.
* Patients who have hepatic and renal parameters within 2X ULN (upper level of normality) at screening.

Exclusion Criteria:

* Patients with a history of hypersensitivity to fluconazole or hLF1-11.
* Patients who have been treated with fluconazole for at least 1 week within the previous 4 weeks.
* Patients with a history of fluconazole-resistant Candida species within 12 weeks.
* Neutropenic patients with neutrophil count below 0.5x10^9/L.
* Patients who are treated with terfenadine, triazolam, cisapride, and ergotamine, which are contraindicated for concomitant use with fluconazole.
* Patients known to have AIDS or who are HIV-positive.
* Females who have a positive pregnancy test at baseline or are capable of child-bearing i.e. without appropriate contraception (chemical or mechanical).
* Patients with suspected candida osteomyelitis, endocarditis, or meningitis.
* Patients who have received an investigational drug within three months prior to the study.
* Patients with a concomitant medical condition, in whom, in the opinion of the Investigator, participation may create an unacceptable risk for the patient.
* Patients considered inappropriate by the PI for enrollment in the study, for any reason.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-01 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Haematology, biochemistry, and microbiological evaluation Adverse event monitoring. | 28 Days

SECONDARY OUTCOMES:
Test of Cure (TOC): Clinical: complete resolution of clinical signs and symptoms or resolution to a point where no further antifungal therapy is judged necessary; and Microbiological: eradication of Candida identified at baseline. | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Professor P.E. Verweij, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- UMC St. Radboud, Nijmegen, Gelderland, Netherlands